CLINICAL TRIAL: NCT03580447
Title: The Effect of Citrus Extract Administration on Markers of Oxidative Stress in Elderly Subjects
Brief Title: The Effect of Citrus Extract on Oxidative Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Yala Stevens, MSc., Maastricht University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 183018
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Elderly
MeSH Terms: interventions — grapefruit seed extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citrus extract (Experimental): During this period participants receive daily citrus extract supplements for four weeks
  Interventions: Dietary Supplement: Citrus extract
- Placebo (Placebo Comparator): During this period participants receive daily maltodextrin supplements for four week
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Citrus extract — Citrus extract
  Arms: Citrus extract
Dietary Supplement: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
This randomized, cross-over, double-blind, placebo-controlled trial aims to determine the effects of daily administration of citrus extract over a period of 4 weeks on markers of oxidative stress in elderly.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Age 70-85 years
* BMI < 30 kg/m2

Exclusion Criteria:

* History or actual status of severe cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological diseases, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol.
* Disease with a life expectancy shorter than 5 years
* Institutionalized (e.g. hospital or nursing home).
* Subjects with abnormalities in haematology which may interfere with the endpoints of the study (to be decided by the principle investigator)
* Use of drugs or hormones within 3 months prior to the start of the study which may interfere with the endpoints of the study (to be decided by the principle investigator)
* Self-admitted Inflammation, (viral) infection (e.g. HIV or hepatitis B)
* Subjects with an autoimmune disease (e.g. Rheumatoid arthritis)
* Subjects with intestinal disorders which may interfere with the endpoints of the study (to be decided by the principle investigator)
* Use of immunosuppressive drugs within 3 months prior to the start of the study
* Use of medication (e.g. NSAIDs), antibiotics or corticosteroids which may interfere with the endpoints of the study (to be decided by the principle investigator)
* Changes in medication that may significantly affect the study outcome (according to the investigator's judgment) within 1 month prior to the start of the study.
* Use of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator) in the 180 days before the study
* Use of (dietary) supplements containing antioxidants, vitamins and minerals
* Smoking
* Weight gain or loss (> 3 kg in the previous 3 months)
* Excessive intake of foods with a high polyphenol concentration
* Use of pre-, pro or synbiotics within 1 month prior to the start of the study
* Blood donation within 1 month prior to the start of the study
* Excessive alcohol consumption (>20 alcoholic consumptions per week)
* History of any side effects towards the intake of flavonoids or citrus fruits

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Oxidative stress | Change from baseline to four weeks supplementation, of each intervention period
  Oxidative stress, as measured by blood biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Ad Masclee, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No